CLINICAL TRIAL: NCT02087020
Title: Debridement, Antibiotics and Implant Retention in Early Periprosthetic Joint Infection: A Retrospective Cohort Study
Acronym: DAIR
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, MD, PhD, Danderyd Hospital
Other Study IDs: DAIR-3
Record Dates: First submitted 2014-03-06; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Direct Infection of Hip- and Knee Arthroplasty
Keywords: Joint Prosthesis; Prosthesis-Related Infections; Joint Diseases; Therapeutic Irrigation; Prostheses and Implants; Arthroplasty Replacement
MeSH Terms: conditions — Prosthesis-Related Infections; Joint Diseases | interventions — Debridement; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Periprosthetic joint infection: Patient treated with 'Debridement, antibiotics and implant retention' for early postoperative periprosthetic joint infection at Danderyd Hospital between 2007-01-01 and 2012-12-01
  Interventions: Procedure: Debridement, antibiotics and implant retention

INTERVENTIONS:
Procedure: Debridement, antibiotics and implant retention — DAIR treatment protocol embodies an extensive surgical debridement and a radical excision of infected tissue. This is followed by exchange of modular components (articulating surfaces of the implant such as the femoral head, acetabular liner in total hip arthroplasty and the tibial insert, the polyethylene meniscus, in total knee arthroplasty). The wound is then copiously irrigated (> 9 litre) with 0.9 % sodium chloride and then closed.

SUMMARY:
Introduction: Periprosthetic joint infection (PJI) is a common cause for reoperation after knee and hip arthroplasty surgery. Debridement, antibiotics and implant retention (DAIR) is recommended in early infections (< 4 weeks) and stable implants. Aims: To define the success rate of DAIR in early infections and to identify predictors for success. Material and methods: In a retrospective cohort study we included patients with hip- or knee arthroplasties reoperated for an early PJI at Danderyd Hospital 2007-2012. Logistic regression analysis was used to identify risk factors affecting success rate. Primary outcome variable was the success of the DAIR treatment. Secondary outcome variable vas risk factors for treatment failure.

ELIGIBILITY:
Inclusion Criteria:

Patients treated with DAIR for early postoperative periprosthetic joint infection after knee- or hip arthroplasty surgery (<4-6 weeks postoperatively) at our institution between 2007-01-01 and 2012-12-01.

Exclusion Criteria:

Chronic or late presenting periprosthetic joint infection (>6 weeks postoperatively), acute hematogenous periprosthetic joint infection, when the periprosthetic joint infection diagnosis criteria according to American Musculoskeletal Infection Society (MSIS) 2011 definition of PJI definitions were not fulfilled and when the initial surgical treatment was with other treatment protocol than DAIR including one-stage revision and two -stage revision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Danderyd Hospital is a university hospital affiliated with the Karolinska Institute and is one of the four emergency hospitals in Stockholm, with a catchment area of approximately 500.000 inhabitants. The index cohort was extracted from the local in-hospital surgery database at the Department of Orthopaedic Surgery using ICD 10 coding and surgical intervention coding for PJI treatment.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Successful treatment | 6 year
  The success rate, in terms of infection eradication without additional surgical methods, of debridement, antibiotics and implant retention in early postoperative periprosthetic joint infection..

SECONDARY OUTCOMES:
Risk factors for treatment failure | 6 year
  Analyze of potential risk factors for treatment failure, age, gender, comorbidities i.e type 1 or 2 diabetes mellitus, renal insufficiency, dementia, systemic inflammatory disease, local or systemic infection, American Society of Anesthesiologists classification, virulence of infecting microbial, hospital stay, typ of arthroplasty, revision arthroplasty, and administration of antibiotics prior to debridement, antibiotics and implant retention treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olof G Skoldenberg, MD,PhD, Principal Investigator — Orthopaedic department, Danderyds hospital; Sebastian S Mukka, MD, Study Chair — Orthopaedic department, Danderyds hospital
Locations (1):
- Danderyd Hospital, Stockholm, Danderyd, Sweden

REFERENCES:
- [Background] Zimmerli W, Trampuz A, Ochsner PE. Prosthetic-joint infections. N Engl J Med. 2004 Oct 14;351(16):1645-54. doi: 10.1056/NEJMra040181. No abstract available. PMID 15483283
- [Derived] Bergkvist M, Mukka SS, Johansson L, Ahl TE, Sayed-Noor AS, Skoldenberg OG, Eisler T. Debridement, antibiotics and implant retention in early periprosthetic joint infection. Hip Int. 2016 Mar-Apr;26(2):138-43. doi: 10.5301/hipint.5000328. Epub 2016 Feb 8. PMID 26868114